CLINICAL TRIAL: NCT07136467
Title: Multi-Country, Cross-sectional Study to Characterize Real World Burden of Disease in Adolescent and Adult Patients With Alopecia Areata, Vitiligo or Hidradenitis Suppurativa (MEASURE AAVitHS)
Brief Title: A Real World Study to Globally Assess Disease Burden in Adolescent and Adult Participants With Alopecia Areata, Vitiligo, or Hidradenitis Suppurativa
Acronym: MEASUREAAVitHS
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H25-663
Record Dates: First submitted 2025-07-31; First posted 2025-08-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non-Segmental Vitiligo (NSV); Alopecia Areata; Hidradenitis Suppurativa
Keywords: Non-Segmental Vitiligo (NSV); Alopecia Areata; Hidradenitis Suppurativa
MeSH Terms: conditions — Alopecia Areata; Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Participants with Vitiligo: Participants with vitiligo will undergo a single-visit data collection per routine clinical practice
- Participants with Alopecia Areata: Participants with alopecia areata will undergo a single-visit data collection per routine clinical practice
- Participants with Hidradenitis Suppurativa: Participants with hidradenitis suppurativa will undergo a single-visit data collection per routine clinical practice

SUMMARY:
This study is to assess the burden of disease in adolescent and adult participants with moderate or severe alopecia areata (AA), non-segmental vitiligo (NSV), or moderate to severe hidradenitis suppurativa (HS) in a large global real-world participant population.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Physician-confirmed diagnosis of non-segmental vitiligo (NSV), moderate to severe Alopecia Areata (AA), or moderate to severe hidradenitis suppurativa (HS)
* Participants Ability to understand study questionnaires, with caregiver support as required for adolescents

Exclusion Criteria:

* Participating in interventional clinical trial(s) at time of study visit (participation in another non-interventional study or registry does not exclude a participant from this study)
* Unable or unwilling to comply with study requirements and PRO collection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and Adult Participants with Alopecia Areata, Vitiligo, or Hidradenitis Suppurativa in Real-World will undergo a single-visit data collection per routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 2795 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Alopecia Areata (AA) symptoms affecting quality of life and daily functioning, assessed by the Alopecia Areata Symptom Impact Scale (AASIS) AA only | Up to Day 1
  AASIS- is a scale assessing the severity of AA-related symptoms on daily functioning. Each item scored on a 0-10 Likert scale, where 0 = not present and 10 = as bad as you can imagine Higher total score = greater impact
Measuring scalp hair loss, assessed by the Severity of Alopecia Tool (SALT) score. AA only | Up to Day 1
  SALT is a Tool developed to quantify AA-related hair loss Total score of 0-100, with 0 = no hair loss, and 100 = complete hair loss
Measuring facial skin depigmentation, assessed by the Facial Vitiligo Area Scoring Index (F-VASI) Vitiligo Only | Up to Day 1
  F-VASI is a quantitative scoring tool used to evaluate the extent and severity of facial vitiligo calculated by multiplying the degree of skin depigmentation of the face
Vitiligo Quality of Life (QOL), assessed by Vitiligo Quality of Life Score (VitiQoL) Vitiligo Only | Up to Day 1
  VitiQoL is a 16-item instrument assessing impact of vitiligo on QoL. 15 items are scored on a 7-point Likert scale, ranging from "not at all" to "all the time". An additional item (not contributing to total score) assesses current severity of condition on a 7-point scale ranging from "no skin involvement" to "most severe case"
Hidradenitis Suppurativa (HS) Quality of Life (QOL), assessed by Dermatology Life Quality Index (DLQI)/Children's Dermatology Life Quality Index (CDLQI) HS only | Up to Day 1
  CDLQI is a10-question index measuring health-related quality of life (HRQoL) over the last 7 days for patients suffering from a skin disease. The DLQI is used in participants aged 16 and over and the CDLQI has been validated from the ages of 4 to 16 years. Each item scored on a 4-point Likert scale, where 0 = not at all/not relevant/question unanswered and 3 = very much. Maximum total score = 30 (highest impact on QoL).
Measuring disease severity, assessed by the International Hidradenitis Suppurativa Severity Scoring System (IHS4) HS only | Up to Day 1
  The IHS4 score is calculated as follows: number of nodules (multiplied by 1) + number of abscesses (multiplied by 2) + number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild, 4 to 10 signifies moderate, and 11 or higher signifies severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (88):
- Argentina (4):
  - Buenos Aires Skin /ID# 277637, Buenos Aires
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC) /ID# 277634, Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 277636, Buenos Aires
  - Instituto de Neumonología y Dermatología /ID# 277635, Buenos Aires
- Canada (5):
  - Alberta Dermatology Consultants /ID# 277187, Edmonton, Alberta
  - Simcoderm Medical And Surgical Dermatology Centre /ID# 276838, Barrie, Ontario
  - DermEffects /ID# 276594, London, Ontario
  - Lynderm Research Inc /ID# 276595, Markham, Ontario
  - York Dermatology Clinic & Research Centre /ID# 276697, Richmond Hill, Ontario
- Dermafit Centrum /ID# 275863, Pilsen, Plzeň Region, Czechia
- North Estonia Medical Centre /ID# 276933, Tallinn, Harju, Estonia
- France (19):
  - Chu Dijon /Id# 277493, Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Régional Universitaire de Besançon - Hôpital Jean Minjoz /ID# 277459, Besançon, Doubs
  - Centre Hospitalier Universitaire de Bordeaux - Groupe Hospitalier Saint-Andre /ID# 277322, Bordeaux, Gironde
  - Centre Hospitalier Régional Universitaire De Tours - Hôpital Trousseau /ID# 277545, Chambray-lès-Tours, Indre-et-Loire
  - Centre Hospitalier de Bretagne Sud /ID# 277559, Lorient, Morbihan
  - Centre Hospitalier Régional Metz Thionville - Hôpital de Mercy /ID# 277792, Metz, Moselle
  - CHU Limoges - Dupuytren 2 /ID# 277323, Limoges, Nouvelle-Aquitaine
  - Médipôle Lyon-Villeurbanne /ID# 277526, Villeurbanne, Rhone
  - Groupe Hospitalier Du Havre - Hôpital Jacques Monod /ID# 277506, Montivilliers, Seine-Maritime
  - Hopital Nord Franche-Comté /ID# 277560, Trévenans, Territoire De Belfort
  - Hôpital d'Instruction des Armées Sainte-Anne /ID# 277458, Toulon, Var
  - Centre Hospitalier Departemental Vendee (Chd Vendee) /ID# 277317, La Roche-sur-Yon, Vendee
  - Centre Hospitalier de Calais /ID# 277320, Calais
  - Cideazur /ID# 277316, Nice
  - Centre De Santé Sabouraud /ID# 278409, Paris
  - Groupe Hospitalier Paris Saint-Joseph /ID# 278270, Paris
  - CHU Rennes - Hôpital PONTCHAILLOU /ID# 277527, Rennes
  - CHU de la reunion /ID# 277318, Saint-Denis
  - Hôpital d'Instruction des Armées Bégin /ID# 278135, Saint-Mandé
- Germany (19):
  - Derma Sana /ID# 279254, Karlsruhe, Baden-Wurttemberg
  - Private Practice - Dr. Virgil Oreste Mihaescu /ID# 279229, Augsburg, Bavaria
  - Hautarztpraxis Hassberge Dr. Boris Bauer /ID# 279272, Haßfurt, Bavaria
  - Dr. Neumann /ID# 279255, Kelheim, Bavaria
  - Dermakulm /Id# 279126, Kulmbach, Bavaria
  - Studienzentrum an der Hase GbR Dr. Weyergraf/Dr. Frick/Thomas Heiber /ID# 279210, Bramsche, Lower Saxony
  - Hautarztliche Gemeinschaftspraxis Dres. med. Petri & Mocklinghoff /ID# 279230, Ahaus, North Rhine-Westphalia
  - Hautarztpraxis Shirin Samimi-Fard & Elena Dippel /ID# 279232, Gladbeck, North Rhine-Westphalia
  - ZENTderma /ID# 279235, Mönchengladbach, North Rhine-Westphalia
  - Private Practice - Dr. Dariusch Mortazawi /ID# 279214, Remscheid, North Rhine-Westphalia
  - Dermatologie Quist-BAG Dres. med. Quist PartG /ID# 279271, Mainz, Rhineland-Palatinate
  - HMS GmbH Zimmer /ID# 279211, Merzig, Saarland
  - Private Practice - Dr. Abdou Zarzour /ID# 279125, Halle, Saxony-Anhalt
  - Private Practice - Dr. Dirk Lange /ID# 279215, Gera, Thuringia
  - MVZ medicum.mittelhessen /ID# 279136, Bad Camberg
  - Hautarztpraxis Dr. Med. Ulrike Wiemers / Dr. Med. Franca Wiemers /ID# 279124, Leipzig
  - Hautarztpraxis Schwelm /ID# 279140, Schwelm
  - Praxis Dehmel / Brand-Opitzer /ID# 279351, Wasserburg A. Inn
  - Dr. med. Nicola Möller & Thomas Kurtenbach GbR Dermatologie im Zentrum /ID# 279137, Wiesbaden
- Greece (2):
  - Tzaneio Prefecture General Hospital of Piraeus /ID# 276881, Piraeus, Attica
  - The University Hospital of Larissa /ID# 277234, Larissa, Larisa
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale S.Anna /ID# 276986, Cona, Ferrara
  - A.O.U. Consorziale Policlinico di Bari /ID# 276857, Bari
- Japan (2):
  - Nagomi Dermatology Clinic /ID# 279997, Ebina-shi, Kanagawa
  - Inokashira Park Skin Clinic /ID# 279276, Mitaka-shi, Tokyo
- Riga 1st Hospital /ID# 276361, Riga, Latvia
- Puerto Rico (3):
  - Dermatologia Borinquen LLC /ID# 276802, Caguas
  - Dr. Samuel Sanchez PSC /ID# 276386, Caguas
  - Clinical Research Puerto Rico /ID# 276801, San Juan
- Romania (7):
  - Institutul Dermato - Estetic /ID# 276296, Bucharest, București
  - Dr. Carol Davila Central Military Emergency University Hospital /ID# 275818, Bucharest, București
  - Spitalul Universitar De Urgență Elias /ID# 275806, Bucharest, București
  - Spitalul Clinic Colentina /ID# 275506, Bucharest, București
  - Spitalul Clinic Colentina /ID# 275817, Bucharest, București
  - Spitalul Clinic Judetean de Urgenta Cluj -Napoca /ID# 276837, Cluj-Napoca, Cluj
  - Spitalul Clinic Județean de Urgențe "Sfântul Spiridon" /ID# 276308, Iași
- South Korea (2):
  - Yonsei University Health System Severance Hospital /ID# 278972, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 278973, Seoul, Seoul Teugbyeolsi
- Hospital Arnau De Vilanova /ID# 276887, Valencia, Spain
- Switzerland (9):
  - Kantonsspital Aarau /ID# 276810, Aarau, Canton of Aargau
  - University Hospital Basel /ID# 276716, Basel Town, Canton of Basel-City
  - Cabinet Dr Damjan Nikolic, Clinique du Seujet /ID# 278467, Geneva, Canton of Geneva
  - Hopitaux Universitaires de Geneve /ID# 277950, Geneva, Canton of Geneva
  - Luzern Kantonsspital /ID# 276813, Lucerne, Canton of Lucerne
  - Praxis Dr. med. Pierre de Viragh /ID# 276855, Zurich, Canton of Zurich
  - Ospedale Regionale Bellinzona E Valli /ID# 277964, Bellinzona, Canton Ticino
  - Studio Medico Dr. Pelloni Francesco /ID# 277948, Lugano, Canton Ticino
  - Inselspital, Universitaetsspital Bern /ID# 276718, Bern
- Taiwan (2):
  - Tri-Service General Hospital /ID# 279761, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 279760, Taoyuan
- United Kingdom (8):
  - University Hospital Lewisham /ID# 279233, London, Greater London
  - Oxford University Hospitals - John Radcliffe Hospital /ID# 279052, Oxford, Oxfordshire
  - Leeds Teaching Hospitals NHS Trust /ID# 278524, Leeds, West Yorkshire
  - Mid Yorkshire Teaching NHS Trust /ID# 279190, Wakefield, West Yorkshire
  - Ulster Hospital - South Eastern Health & Social Care Trust /ID# 279191, Belfast
  - Cardiff and Vale UHB /ID# 278856, Cardiff
  - Walsall Manor Hospital /ID# 279240, Walsall
  - New Cross Hospital /ID# 279202, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H25-663